CLINICAL TRIAL: NCT04285528
Title: Intravenous Sedation and Analgesia Using Propofol, Fentanyl and Ketamine (PFK) Versus General Anesthesia in Minor Urological Procedures.
Brief Title: Sedation and Analgesia Using PFK Versus General Anesthesia in Urological Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Abdelkarim Saleh AlOweidi, Principal investigator, University of Jordan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 67/2019/1166
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia; Urologic Diseases
Keywords: General anesthesia; Sedation; Propofol; Fentanyl; Ketamine; Hypotension
MeSH Terms: conditions — Urologic Diseases; Hypotension | interventions — Propofol; Ketamine; Fentanyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- General Anesthesia (Experimental): The first group which will undergo general anesthesia, will be anesthetized using Fentanyl (2 mcg per kg) and Propofol (1-2 mg per kg). Laryngeal mask airway will be inserted afterwards.
  Interventions: Drug: General anesthetia Fentanyl and Propofol
- PFK group (Experimental): The second group will undergo intravenous sedation and analgesia by using a mixture of Fentanyl, Propofol and Ketamine (PFK mixture). The mixture consists of 100 mcg Fentanyl, 100 mg Propofol, 100 mg of Ketamine. In addition, 40 mg of Lidocaine will be added, this aims to reduce the pain on injection caused by Propofol. Moreover, 4 ml of water for injection will be added to the mixture.
  Interventions: Combination Product: PFK

INTERVENTIONS:
Drug: General anesthetia Fentanyl and Propofol — Patients were anesthetized using Fentanyl (2 mcg per kg) and Propofol (1-2 mg per kg). Proper classic laryngeal mask airway was inserted afterwards.
  Other Names: GA
  Arms: General Anesthesia
Combination Product: PFK — A mixture of 5 mcg/ml of Fentanyl, 5 mg/ml of Propofol, and 5 mg/ml of Ketamine was used. Each patient received an initial dose of 0.5 mg/kg from the solution, then after waiting for 60 seconds, another 0.5 mg/kg were given. Maintenance was given as boluses of 0.2- 0.33 mg/kg every three to five minutes. No Laryngeal mask airway nor endotracheal tube were inserted, and the patients were breathing spontaneously through a simple face mask on a support of 3 L/min O2.
  Other Names: propofol-ketamine-fentanyl (PFK) mixture; the mixture of propofol, ketamine, fentanyl, with lidocaine
  Arms: PFK group

SUMMARY:
Anesthesia in urological surgeries might constitute a great challenge to anesthesiologists. Especially that a great proportion of these patients are elderly with a lot of comorbidities. This put these patients at the risk of developing medical adverse events after being anesthetized by general anesthesia. The aim of this study is to compare between intravenous sedation with analgesia versus general anesthesia in patients undergoing urological surgical procedures.

DETAILED DESCRIPTION:
Anesthesia in urological surgeries might constitute a great challenge to anesthesiologists. Especially that a great proportion of these patients are elderly with a lot of comorbidities. This put these patients at the risk of developing medical adverse events after being anesthetized by general anesthesia. The aim of this study is to compare between intravenous sedation with analgesia versus general anesthesia in patients undergoing urological surgical procedures.

The first group which underwent general anesthesia, was anesthetized using Fentanyl (2 mcg per kg) and Propofol (1-2 mg per kg). Laryngeal mask airway was then inserted.

The second group underwent intravenous sedation and analgesia by using a mixture of Fentanyl, Propofol and Ketamine (PFK mixture). The mixture consists of 100 mcg Fentanyl, 100 mg Propofol, 100 mg of Ketamine. In addition, 40 mg of Lidocaine were added, this aimed to reduce the pain on injection caused by Propofol. Moreover, 4 ml of water of injection were added to the mixture. This resulted in a mixture of 5 mcg/ml of Fentanyl, 5 mg/ml of Propofol, and 5 mg/ml of Ketamine. By this, each ml of the mixture contained 10 mg (ketamine and propofol) + 5 mcg fentanyl. Each patient received an initial dose of 0.5 mg/kg from the solution, then after waiting for 60 seconds, another 0.5 mg/kg were given. Maintenance was given as boluses of 0.2- 0.33 mg/kg every three to five minutes. No laryngeal mask airway nor endotracheal tube were inserted, and the patients were breathing spontaneously through a simple face mask on support of 3 L/min O2.

ELIGIBILITY:
Inclusion Criteria:

* patients above the age of 30 years
* patients who were admitted for minor urological surgeries under the care of urology team. Minor urological procedures, included cystoscopy, trans-urethral resection of tumor (TURT), uretroscopy, double J insertion, and double J removal.

Exclusion Criteria:

* patient refusal.
* urgent and emergency cases, which were not elective procedures.
* Surgeries that were expected to take a long duration (more than 1.5 hour).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure stability | 45 minutes
  the investigators recorded the changes in blood pressure after induction of anesthesia

SECONDARY OUTCOMES:
Hypoxia | 45 minutes
  the investigators recorded any episodes of transient reduction of oxygen saturation.
nausea and vomiting | 2 hours
  The investigators recorded the occurrence of nausea and vomiting till the discharge of the patients from post anesthesia care unit (PACU).

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White PF, Kehlet H, Neal JM, Schricker T, Carr DB, Carli F; Fast-Track Surgery Study Group. The role of the anesthesiologist in fast-track surgery: from multimodal analgesia to perioperative medical care. Anesth Analg. 2007 Jun;104(6):1380-96, table of contents. doi: 10.1213/01.ane.0000263034.96885.e1. PMID 17513630
- [Background] Jalili M, Bahreini M, Doosti-Irani A, Masoomi R, Arbab M, Mirfazaelian H. Ketamine-propofol combination (ketofol) vs propofol for procedural sedation and analgesia: systematic review and meta-analysis. Am J Emerg Med. 2016 Mar;34(3):558-69. doi: 10.1016/j.ajem.2015.12.074. Epub 2015 Dec 29. PMID 26809929
- [Background] Ferguson I, Bell A, Treston G, New L, Ding M, Holdgate A. Propofol or Ketofol for Procedural Sedation and Analgesia in Emergency Medicine-The POKER Study: A Randomized Double-Blind Clinical Trial. Ann Emerg Med. 2016 Nov;68(5):574-582.e1. doi: 10.1016/j.annemergmed.2016.05.024. Epub 2016 Jul 22. PMID 27460905
- [Background] David H, Shipp J. A randomized controlled trial of ketamine/propofol versus propofol alone for emergency department procedural sedation. Ann Emerg Med. 2011 May;57(5):435-41. doi: 10.1016/j.annemergmed.2010.11.025. Epub 2011 Jan 21. PMID 21256626
- [Background] Morrison K, Herbst K, Corbett S, Herndon CD. Pain management practice patterns for common pediatric urology procedures. Urology. 2014 Jan;83(1):206-10. doi: 10.1016/j.urology.2013.08.041. Epub 2013 Oct 16. PMID 24139358
- [Background] Borland ML, Bergesio R, Pascoe EM, Turner S, Woodger S. Intranasal fentanyl is an equivalent analgesic to oral morphine in paediatric burns patients for dressing changes: a randomised double blind crossover study. Burns. 2005 Nov;31(7):831-7. doi: 10.1016/j.burns.2005.05.001. Epub 2005 Jul 6. PMID 16005154
- [Background] Tosun Z, Aksu R, Guler G, Esmaoglu A, Akin A, Aslan D, Boyaci A. Propofol-ketamine vs propofol-fentanyl for sedation during pediatric upper gastrointestinal endoscopy. Paediatr Anaesth. 2007 Oct;17(10):983-8. doi: 10.1111/j.1460-9592.2007.02206.x. PMID 17767636
- [Background] Singh Bajwa SJ, Bajwa SK, Kaur J. Comparison of two drug combinations in total intravenous anesthesia: Propofol-ketamine and propofol-fentanyl. Saudi J Anaesth. 2010 May;4(2):72-9. doi: 10.4103/1658-354X.65132. PMID 20927266
- [Background] Kushikata T, Yatsu Y, Kubota T, Matsuki A. [Total intravenous anesthesia with propofol, ketamine, and fentanyl (PFK) for a patient with mitochondrial myopathy]. Masui. 2004 Feb;53(2):178-80. Japanese. PMID 15011427
- [Background] Kakinohana M, Saitoh T, Kakinohana O, Okuda Y. [A case of total intravenous anesthesia with propofol, fentanyl and ketamine for lateral segmentectomy of the liver under pringle maneuver]. Masui. 1999 May;48(5):523-7. Japanese. PMID 10380509
- [Background] Tokumine J, Iha H, Okuda Y, Shimabukuro T, Shimabukuro T, Ishigaki K, Nakamura S, Takara I. Appropriate method of administration of propofol, fentanyl, and ketamine for patient-controlled sedation and analgesia during extracorporeal shock-wave lithotripsy. J Anesth. 2000 Apr 25;14(2):68-72. doi: 10.1007/s005400050069. PMID 14564593
- [Background] Lonjaret L, Lairez O, Minville V, Geeraerts T. Optimal perioperative management of arterial blood pressure. Integr Blood Press Control. 2014 Sep 12;7:49-59. doi: 10.2147/IBPC.S45292. eCollection 2014. PMID 25278775
- [Background] Atashkhoyi S, Negargar S, Hatami-Marandi P. Effects of the addition of low-dose ketamine to propofol-fentanyl anaesthesia during diagnostic gynaecological laparoscopy. Eur J Obstet Gynecol Reprod Biol. 2013 Sep;170(1):247-50. doi: 10.1016/j.ejogrb.2013.06.026. Epub 2013 Jul 17. PMID 23870189
- [Background] Hayakawa-Fujii Y, Takada M, Ohta S, Dohi S. Hemodynamic stability during induction of anesthesia and tracheal intubation with propofol plus fentanyl, ketamine, and fentanyl-ketamine. J Anesth. 2001;15(4):191-6. doi: 10.1007/s005400170001. PMID 14569434
- [Background] Tang YY, Lin XM, Huang W, Jiang XQ. Addition of low-dose ketamine to propofol-fentanyl sedation for gynecologic diagnostic laparoscopy: randomized controlled trial. J Minim Invasive Gynecol. 2010 May-Jun;17(3):325-30. doi: 10.1016/j.jmig.2010.01.017. PMID 20417423
- [Background] Saadawy I, Ertok E, Boker A. Painless injection of propofol: pretreatment with ketamine vs thiopental, meperidine, and lidocaine. Middle East J Anaesthesiol. 2007 Oct;19(3):631-44. PMID 18044291
- [Background] Erden IA, Pamuk AG, Akinci SB, Koseoglu A, Aypar U. Comparison of propofol-fentanyl with propofol-fentanyl-ketamine combination in pediatric patients undergoing interventional radiology procedures. Paediatr Anaesth. 2009 May;19(5):500-6. doi: 10.1111/j.1460-9592.2009.02971.x. PMID 19453582
- [Background] Sakai T, Mi WD, Komoda Y, Kudo T, Kudo M, Matsuki A. [Clinical indication of propofol for pediatric patients--pharmacokinetics of propofol and ketamine during and after total intravenous anesthesia with propofol, fentanyl and ketamine (PFK) in a neonate]. Masui. 1998 Mar;47(3):314-7. Japanese. PMID 9560543
- [Background] Childers CP, Maggard-Gibbons M. Understanding Costs of Care in the Operating Room. JAMA Surg. 2018 Apr 18;153(4):e176233. doi: 10.1001/jamasurg.2017.6233. Epub 2018 Apr 18. PMID 29490366
- [Background] Berning V, Laupheimer M, Nubling M, Heidegger T. Influence of quality of recovery on patient satisfaction with anaesthesia and surgery: a prospective observational cohort study. Anaesthesia. 2017 Sep;72(9):1088-1096. doi: 10.1111/anae.13906. Epub 2017 May 16. PMID 28510285
- [Background] Onaka M, Akatsuka M, Takayama R, Mori H, Yamamoto H. [Electroencephalographic characteristics during maintenance and emergence from propofol-ketamine-fentanyl anesthesia]. Masui. 2001 Mar;50(3):265-9. Japanese. PMID 11296437